CLINICAL TRIAL: NCT00934635
Title: The "Therapeutic Window" of the "Atypical" Antipsychotic Paliperidone Extended Release (ER)-A Positron Emission Tomography Study With [18F]Fallypride as the Radiotracer
Brief Title: A Positron-Emission-Tomography (PET) Study to Measure the Blockade of Dopamine Receptors (D2) in Specific Areas of the Brain in Relation to the Plasma Concentrations of Paliperidone Extended Release (ER) and Oral Risperidone in Schizophrenia Patients and Healthy Controls
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag G.m.b.H (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015277
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Results first posted 2011-01-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-01

CONDITIONS: Schizophrenia
Keywords: D2-receptor occupancy; Antipsychotic drugs; Paliperidone ER, Oral risperidone; Dopamine; Fallypride; Plasma concentration; Therapeutic window, Healthy controls
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate; Risperidone; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- 002 (Active Comparator): Paliperidone ER 9 mg tablet once a day followed by PET scan in approximately 2 hours
  Interventions: Drug: Paliperidone ER
- 003 (Active Comparator): Oral risperidone 4 mg tablet once a day followed by PET scan in approximately 2 hours
  Interventions: Drug: Oral risperidone
- 004 (Active Comparator): Oral risperidone 6 mg tablet once a day followed by PET scan in approximately 2 hours
  Interventions: Drug: Oral risperidone
- 005 (Active Comparator): Paliperidone ER 6 mg tablet once a day followed by PET scan in approximately 24 hours
  Interventions: Drug: Paliperidone ER
- 006 (Active Comparator): Paliperidone ER 9 mg tablet once a day followed by PET scan in approximately 24 hours
  Interventions: Drug: Paliperidone ER
- 007 (Active Comparator): Oral risperidone 4 mg tablet once a day followed by PET scan in approximately 24 hours
  Interventions: Drug: Oral risperidone
- 008 (Active Comparator): Oral risperidone 6 mg tablet once a day followed by PET scan in approximately 24 hours
  Interventions: Drug: Oral risperidone
- 009 (Other): PET Scan PET Scan
  Interventions: Other: PET Scan
- 001 (Active Comparator): Paliperidone ER 6 mg tablet once a day followed by PET scan in approximately 2 hours
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — 9 mg tablet once a day followed by PET scan in approximately 2 hours
  Arms: 002
Drug: Oral risperidone — 6 mg tablet once a day followed by PET scan in approximately 2 hours
  Arms: 004
Other: PET Scan — PET Scan
  Arms: 009
Drug: Oral risperidone — 4 mg tablet once a day followed by PET scan in approximately 24 hours
  Arms: 007
Drug: Oral risperidone — 4 mg tablet once a day followed by PET scan in approximately 2 hours
  Arms: 003
Drug: Paliperidone ER — 6 mg tablet once a day followed by PET scan in approximately 2 hours
  Arms: 001
Drug: Paliperidone ER — 6 mg tablet once a day followed by PET scan in approximately 24 hours
  Arms: 005
Drug: Oral risperidone — 6 mg tablet once a day followed by PET scan in approximately 24 hours
  Arms: 008
Drug: Paliperidone ER — 9 mg tablet once a day followed by PET scan in approximately 24 hours
  Arms: 006

SUMMARY:
The primary objective of this study is to compare the effect of two different antipsychotic compounds which are used in the treatment of schizophrenia (paliperidone ER and risperidone) at their target sites in two specific areas of the brain in patients with schizophrenia. A specialized X-ray known as Positron Emission Tomography (PET) Imaging is used to assess the areas of the brain targeted by both compounds.

DETAILED DESCRIPTION:
This is an open-label (all people involved know the identity of the intervention), non-randomized (patients are assigned to treatment groups), phase IV, monocentric (at one single study site) interventional study evaluating the blocking effects two different doses of paliperidone ER and oral risperidone have on the dopamine D2 receptors in the brain of subchronic patients with schizophrenia. Dopamine is a substance produced and released in the brain. Research indicates that dopamine levels are elevated in some areas of the brain in acute schizophrenia psychosis. Antipsychotic medications like risperidone and paliperidone ER are used to treat psychosis by blocking the dopamine receptors. Fallypride is a radioactive tracer (a drug that emits radioactivity) that binds to the dopamine receptors in the brain much the same as antipsychotic medications. It competes with the antipsychotic compounds at the binding sites and is used when performing a specialized x-ray known as Positron Emission Tomography (PET) Imaging. After a patient receives Fallypride, it temporally binds to specific target areas in the brain and emits a brief and harmless radioactive signal that is detected by the PET Scanner. Since paliperidone ER and risperidone compete with Fallypride at the same target sites, the signal will differ according to the binding effect of the compound. This technique provides an image showing the direct effect medication has on the human brain and allows for comparisons of the effects of different medications to be made. As this effect will fluctuate depending on the concentration of the drug in the blood, during this study, PET measurements will be correlated with the blood levels sampled. Patients will receive either paliperidone ER (6 patients with 6 mg per day, 6 patients with 9 mg per day) or oral risperidone (6 patients with 4 mg per day, 6 patients with 6 mg per day). The primary objective of this study is to compare the blocking effects each medication has on the dopamine D2 receptors at different time points (shortly after taking medication and 24 hours after taking medication) correlated with blood levels of the medication. The study consists of 3 visits on 3 consecutive days. Blood levels will be assessed for treatment groups 1 to 4 on day 2 and day 3 and for groups 5 to 8 on day 3 (according to the last intake of study medication). PET-Scans will be assessed for every group on day 3. Group 1 to 4 consists of patients whose PET Scan will be assessed approximately 2 hours after taking medication (group 1 receives paliperidone ER 6 mg, group 2 receives paliperidone ER 9 mg, group 3 receives risperidone 4 mg, group 4 receives risperidone 6 mg). Group 5 to 8 consists of patients whose PET Scan will be assessed approximately 24 hours after taking medication (group 5 receives paliperidone ER 6 mg, group 6 receives paliperidone ER 9 mg, group 7 receives risperidone 4 mg, group 8 receives risperidone 6 mg). Adverse Events (AE's) will be assessed as reported spontaneously throughout the trial. The dose of antipsychotic medication will represent the most frequent dose used in post acute treatment of schizophrenia. A group of healthy volunteers (group 9) will serve as a control group to measure fallypride dopamine D2- receptor occupancies under normal circumstances, in patients not affected by schizophrenia. Patients will receive the same dosage throughout the study as prescribed prior to the start of the study either paliperidone ER 6 mg tablet once daily or 9 mg tablet once daily or risperidone 4 mg tablet once daily or 6 mg daily (two 3 mg tablets).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria
* Patients with a specified severity of the disease (Clinical Global Impression Scale of Severity (CGI-S) range of > 2 < 5)
* Patients must be on antipsychotic medication with either paliperidone ER or oral risperidone in monotherapy for at least two weeks and must be at least five days on a stable dose of either paliperidone ER 6 mg or 9 mg or oral risperidone 4 mg or 6 mg once daily
* Female patients of childbearing potential must have a negative human chorionic gonadotropin urine pregnancy test (ß-HCG) at visit 1 or must be postmenopausal for at least 1 year, surgically sterile, abstinent, or, if sexually active, agree to practice an effective method of birth control before entry, throughout the study and at least one month after study end
* Healthy control volunteers must be off all standard prescription drug therapy, over the counter compounds (OTC) and recreational substances/drugs for at least one week prior to participation in the study
* Female volunteers of childbearing potential must have a negative ß -HCG pregnancy test at visit 1 or be postmenopausal for at least 1 year, surgically sterile, abstinent, or, if sexually active, agree to practice an effective method of birth control before entry, throughout the study and at least one month after the study end
* Patients and volunteers must be able to read, understand and sign the Institutional Review Board approved informed consent form

Exclusion Criteria:

* Patients: Any depot neuroleptic medication (long acting injectables) in the last three months
* Any antipsychotic compound, antidepressant, antiepileptic ("mood stabilizers"), lithium, anticholinergic within 2 weeks prior to study
* Any psychopharmacologically active medication (except benzodiazepines, paracetamol and zopiclone as rescue medication) taken within the trial
* Physical and psychological conditions that interfere with the study procedures, or could influence the study results, or could endanger the patient during the study
* Alcohol and/or drug abuse four weeks prior to study start (patients with alcohol or drug abuse as defined by the DSM-IV criteria can participate if free of their of abuse for at least four weeks)
* Clinically relevant laboratory abnormality
* Pregnant or breast feeding patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag G.m.b.H. Clinical Trial, Study Director — Janssen-Cilag G.m.b.H
Locations (1):
- Aachen, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone ER 6 mg Tablet Followed by PET Scan in 2 Hours: Paliperidone ER 6 mg tablet once a day (for 2 days) followed by PET scan in approximately 2 hours
- Paliperidone ER 9 mg Tablet Followed by PET Scan in 2 Hours: Paliperidone ER 9 mg tablet once a day (for 2 days) followed by PET scan in approximately 2 hours
- Oral Risperidone 4 mg Tablet Followed by PET Scan in 2 Hours: Oral risperidone 4 mg tablet once a day (for 2 days) followed by PET scan in approximately 2 hours
- Oral Risperidone 6 mg Tablet Followed by PET Scan in 2 Hours: Oral risperidone 6 mg tablet once a day (for 2 days)followed by PET scan in approximately 2 hours
- Paliperidone ER 6 mg Tablet Followed by PET Scan in 24 Hours: Paliperidone ER 6 mg tablet once a day (1 day intake, one day off) followed by PET scan in 24 hours
- Paliperidone ER 9 mg Tablet Followed by PET Scan in 24 Hours: Paliperidone ER 9 mg tablet once a day (1 day intake, 1 day off) followed by PET scan in approximately 24 hours
- Oral Risperidone 4 mg Tablet Followed by PET Scan in 24 Hours: Oral risperidone 4 mg tablet once a day (1 day intake; 1 day off) followed by PET scan in approximately 24 hours
- Oral Risperidone 6 mg Tablet Followed by PET Scan in 24 Hours: Oral risperidone 6 mg tablet once a day (1 day intake; 1 day off) followed by PET scan in approximately 24 hours
- Control: PET Scan Control
Period: Overall Study
Arm/Group | Paliperidone ER 6 mg Tablet Followed by PET Scan in 2 Hours | Paliperidone ER 9 mg Tablet Followed by PET Scan in 2 Hours | Oral Risperidone 4 mg Tablet Followed by PET Scan in 2 Hours | Oral Risperidone 6 mg Tablet Followed by PET Scan in 2 Hours | Paliperidone ER 6 mg Tablet Followed by PET Scan in 24 Hours | Paliperidone ER 9 mg Tablet Followed by PET Scan in 24 Hours | Oral Risperidone 4 mg Tablet Followed by PET Scan in 24 Hours | Oral Risperidone 6 mg Tablet Followed by PET Scan in 24 Hours | Control
Started | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paliperidone ER 6 mg Tablet Followed by PET Scan in 2 Hours | Paliperidone ER 9 mg Tablet Followed by PET Scan in 2 Hours | Oral Risperidone 4 mg Tablet Followed by PET Scan in 2 Hours | Oral Risperidone 6 mg Tablet Followed by PET Scan in 2 Hours | Paliperidone ER 6 mg Tablet Followed by PET Scan in 24 Hours | Paliperidone ER 9 mg Tablet Followed by PET Scan in 24 Hours | Oral Risperidone 4 mg Tablet Followed by PET Scan in 24 Hours | Oral Risperidone 6 mg Tablet Followed by PET Scan in 24 Hours | Control | Total
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 |  |  |  |  |  |  | 0 | 0
  Between 18 and 65 years |  | 1 |  |  |  |  |  |  | 1 | 2
  >=65 years |  | 0 |  |  |  |  |  |  | 0 | 0
Age, Customized [Number; unit: years]
  27 years of age |  | 1 (NA) |  |  |  |  |  |  | 0 (NA) | 1
  19 years of age |  | 0 |  |  |  |  |  |  | 1 | 1
Gender [Number; unit: participants]
  Female |  | 0 |  |  |  |  |  |  | 1 | 1
  Male |  | 1 |  |  |  |  |  |  | 0 | 1
Region of Enrollment [Number; unit: participants]
  Germany |  | 1 |  |  |  |  |  |  | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Paliperidone or Risperidone Dopamine D2 Receptor Occupancies
Time Frame: Visit 3 (on day 3)
Population: PET imaging data were not submitted for further analysis. D2-receptor occupancies could not be calculated due to the low number of subjects in the healthy control group.
Measure: Number; unit: percentage
Arm/Group | Paliperidone ER 6 mg Tablet Followed by PET Scan in 2 Hours | Paliperidone ER 9 mg Tablet Followed by PET Scan in 2 Hours | Oral Risperidone 4 mg Tablet Followed by PET Scan in 2 Hours | Oral Risperidone 6 mg Tablet Followed by PET Scan in 2 Hours | Paliperidone ER 6 mg Tablet Followed by PET Scan in 24 Hours | Paliperidone ER 9 mg Tablet Followed by PET Scan in 24 Hours | Oral Risperidone 4 mg Tablet Followed by PET Scan in 24 Hours | Oral Risperidone 6 mg Tablet Followed by PET Scan in 24 Hours | Control
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
percentage |  | 0 |  |  |  |  |  |  | 0

2. Secondary Outcome: Plasma Concentrations of Paliperidone and Risperidone
Description: No measures available due to early termination of trial
Time Frame: Measurement of plasma concentration at Visit 3 (day 3)
Reporting Status: Not Posted
Measure: Number

3. Secondary Outcome: Assessment of the Ratio of Dopamine D2-receptor Occupancies in Two Different Areas of the Brain
Description: No measures available due to early termination of trial
Time Frame: Analysis of PET scans at Visit 3 (day 3)
Reporting Status: Not Posted
Measure: Number

ADVERSE EVENTS:
Arm/Group | Paliperidone ER 6 mg Tablet Followed by PET Scan in 2 Hours | Paliperidone ER 9 mg Tablet Followed by PET Scan in 2 Hours | Oral Risperidone 4 mg Tablet Followed by PET Scan in 2 Hours | Oral Risperidone 6 mg Tablet Followed by PET Scan in 2 Hours | Paliperidone ER 6 mg Tablet Followed by PET Scan in 24 Hours | Paliperidone ER 9 mg Tablet Followed by PET Scan in 24 Hours | Oral Risperidone 4 mg Tablet Followed by PET Scan in 24 Hours | Oral Risperidone 6 mg Tablet Followed by PET Scan in 24 Hours | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paliperidone ER 6 mg Tablet Followed by PET Scan in 2 Hours (N=0) | Paliperidone ER 9 mg Tablet Followed by PET Scan in 2 Hours (N=1) | Oral Risperidone 4 mg Tablet Followed by PET Scan in 2 Hours (N=0) | Oral Risperidone 6 mg Tablet Followed by PET Scan in 2 Hours (N=0) | Paliperidone ER 6 mg Tablet Followed by PET Scan in 24 Hours (N=0) | Paliperidone ER 9 mg Tablet Followed by PET Scan in 24 Hours (N=0) | Oral Risperidone 4 mg Tablet Followed by PET Scan in 24 Hours (N=0) | Oral Risperidone 6 mg Tablet Followed by PET Scan in 24 Hours (N=0) | Control (N=1)
Exacerbation of schizophrenic symptoms (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — 13 days after patient completed study a SAE report indicated exacerbation of symptoms after illegal drug intake.He was transferred to locked ward, switched to clozapine and symptoms resolved without sequel.SAE classified unrelated to study medication

LIMITATIONS AND CAVEATS:
Two subjects enrolled, both completed study per protocol. Study was prematurely terminated, data obtained were not submitted to further statistical analysis and will not be applicable for scientific analysis due to the low number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study data will be coordinated by the Sponsor, but written by the Investigator.

The Medical Institution will not be entitled to publish any data unless the Sponsor has received the manuscript within 3 months after the Clinical Study Report for review (within 30 days) to ensure that the publication does not reveal secret information. If the Sponsor suggests changes, these changes must be incorporated unless they compromise the scientific nature of the publication.